CLINICAL TRIAL: NCT07333040
Title: Hemorrhoidectomy, Energy-Based, and Laser Outcomes in Grade III Hemorrhoids: A Prospective, Multicenter, Preference-Based Comparative Study
Brief Title: HELO Trial: Energy-Based Therapies vs. Conventional Hemorrhoidectomy for Grade III Hemorrhoids
Acronym: HELO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Taiwan Colorectal Action Research, TCAR (Unknown); Chang Gung Memorial Hospital, Keelung (Unknown); Jen-Ai Hospital Institutional Review Board (Industry); New Taipei City Hospital (Other)
Responsible Party: Principal Investigator, I-Li Lai, MD, Assistant Professor, Chang Gung Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202501172A3
Record Dates: First submitted 2026-01-01; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Hemorrhoids Third Degree; Internal Hemorrhoids; Mixed Hemorrhoids
Keywords: Laser Hemorrhoidoplasty; Hemorrhoid Energy Therapy; Postoperative Pain; Minimally Invasive Surgery; Hemorrhoidectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Due to the distinct physical nature of the surgical interventions (conventional excision vs. energy-based ablation), blinding of participants and care providers is not feasible. To minimize detection bias, the determination of recurrence and the need for re-intervention (secondary endpoint) will be adjudicated by an independent committee blinded to the treatment allocation. Additionally, data regarding patient-reported outcomes (pain, HDSS) will be collected by research staff who are not involved in the surgical procedures.
Who Masked: Outcomes Assessor
Masking Description: Due to the distinct physical nature of the surgical interventions (conventional excision vs. energy-based ablation), blinding of participants and care providers is not feasible. To minimize detection bias, the determination of recurrence and the need for re-intervention (secondary endpoint) will be adjudicated by an independent committee blinded to the treatment allocation. Additionally, data regarding patient-reported outcomes (pain, HDSS) will be collected by research staff who are not involved in the surgical procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laser Hemorrhoidoplasty (LHP) (Experimental): 1470nm or 980nm diode laser ablation
  Interventions: Procedure: Laser Hemorrhoidoplasty (LHP)
- Hemorrhoid Energy Therapy (HET) (Experimental): Bipolar radiofrequency coagulation using HET™ system
  Interventions: Procedure: Hemorrhoid Energy Therapy (HET)
- Conventional Hemorrhoidectomy (Active Comparator): Standard closed excisional hemorrhoidectomy
  Interventions: Procedure: Ferguson Hemorrhoidectomy

INTERVENTIONS:
Procedure: Laser Hemorrhoidoplasty (LHP) — 1470nm or 980nm diode laser ablation
  Arms: Laser Hemorrhoidoplasty (LHP)
Procedure: Hemorrhoid Energy Therapy (HET) — Bipolar radiofrequency coagulation using HET™ system
  Arms: Hemorrhoid Energy Therapy (HET)
Procedure: Ferguson Hemorrhoidectomy — Standard closed excisional hemorrhoidectomy
  Arms: Conventional Hemorrhoidectomy

SUMMARY:
This prospective, multicenter study compares the efficacy and functional outcomes of three surgical treatments for symptomatic Goligher Grade III internal hemorrhoids: Laser Hemorrhoidoplasty (LHP), Hemorrhoid Energy Therapy (HET), and conventional closed hemorrhoidectomy (Ferguson technique). Due to strong patient preferences in hemorrhoidal surgery, this study utilizes a pragmatic, preference-tolerant design. Eligible patients will undergo standardized counseling and select their preferred treatment arm. The study aims to evaluate whether minimally invasive energy-based therapies offer superior postoperative pain relief and faster functional recovery compared to conventional hemorrhoidectomy

DETAILED DESCRIPTION:
This prospective, multicenter trial aims to evaluate and optimize the surgical management of Goligher Grade III internal hemorrhoids. While conventional excisional hemorrhoidectomy (Ferguson technique) remains the gold standard, it is associated with significant postoperative pain and prolonged recovery. Emerging energy-based therapies, specifically Laser Hemorrhoidoplasty (LHP) and Hemorrhoid Energy Therapy (HET), offer potential advantages but their comparative efficacy remains understudied.

The study employs a pragmatic, preference-based design to reflect real-world clinical decision-making. Eligible participants will receive standardized counseling regarding three treatment options: (1) LHP, (2) HET, and (3) Conventional Hemorrhoidectomy, and will be assigned to their preferred treatment arm. To mitigate selection bias, propensity score overlap weighting (PSOW) will be utilized in the statistical analysis.

The primary objective is to compare the postoperative pain trajectory (assessed by the Area Under the Curve of NRS pain scores from Day 1 to Day 14) and the time to functional recovery among the three groups. Secondary objectives include the assessment of 12-month recurrence rates, symptom severity (HDSS), quality of life (Short Health Scale), and postoperative complications. Recurrence outcomes will be adjudicated by an independent blinded committee to minimize detection bias.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Goligher Grade III internal hemorrhoids.
* Symptomatic with HDSS score >= 5.
* Age 18-75 years.
* Fit for general anesthesia or sedation.
* Able to provide informed consent.
* Agree to pre-operative photo documentation.

Exclusion Criteria:

* Other anorectal diseases (fistula, abscess, IBD, malignancy).
* Prior anorectal surgery within 6 months.
* Pregnancy or lactation.
* Contraindications to anesthesia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Time to Functional Recovery | Up to 1 month post-operation
  Days to return to work or normal daily activities.
Post-operative Pain Trajectory (Area Under the Curve) | Post-operative Day 1 to Day 14
  Assessed using Numeric Rating Scale (0-10). Calculated as Area Under the Curve (AUC).

SECONDARY OUTCOMES:
Recurrence Rate | 12 months post-operation
  Defined as the recurrence of prolapse or bleeding requiring medical or surgical re-intervention, or deterioration in HDSS score beyond a prespecified threshold. To ensure objectivity, these events will be adjudicated by an independent committee blinded to the treatment allocation.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Linkou Branch, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Oostendorp JY, Dekker L, van Dieren S, Veldkamp R, Bemelman WA, Han-Geurts IJM; HollAND Study Group. Comparison of Rubber Band Ligation and Hemorrhoidectomy in Patients With Symptomatic Hemorrhoids Grade III: A Multicenter, Open-Label, Randomized Controlled Noninferiority Trial. Dis Colon Rectum. 2025 May 1;68(5):572-583. doi: 10.1097/DCR.0000000000003679. Epub 2025 Feb 14. PMID 39952268
- [Background] Gambardella C, Brusciano L, Brillantino A, Parisi S, Lucido FS, Del Genio G, Tolone S, Allaria A, Di Saverio S, Pizza F, Sturiale A, Docimo L. Mid-term efficacy and postoperative wound management of laser hemorrhoidoplasty (LHP) vs conventional excisional hemorrhoidectomy in grade III hemorrhoidal disease: the twisting trend. Langenbecks Arch Surg. 2023 Apr 5;408(1):140. doi: 10.1007/s00423-023-02879-4. PMID 37020091
- [Background] Hawkins AT, Davis BR, Bhama AR, Fang SH, Dawes AJ, Feingold DL, Lightner AL, Paquette IM; Clinical Practice Guidelines Committee of the American Society of Colon and Rectal Surgeons. The American Society of Colon and Rectal Surgeons Clinical Practice Guidelines for the Management of Hemorrhoids. Dis Colon Rectum. 2024 May 1;67(5):614-623. doi: 10.1097/DCR.0000000000003276. Epub 2024 Jan 31. No abstract available. PMID 38294832
- [Background] Giuliani A, Romano L, Necozione S, Cofini V, Di Donato G, Schietroma M, Carlei F; EMODART3 Study Group. Excisional Hemorrhoidectomy Versus Dearterialization With Mucopexy for the Treatment of Grade III Hemorrhoidal Disease: The EMODART3 Multicenter Study. Dis Colon Rectum. 2023 Dec 1;66(12):e1254-e1263. doi: 10.1097/DCR.0000000000002885. Epub 2023 Aug 24. PMID 37616177